CLINICAL TRIAL: NCT03452345
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center, Phase 3 Study to Evaluate the Efficacy and Safety of MEDOTIXN® in Subject With Benign Masseteric Hypertrophy
Brief Title: MEDITOXIN® Treatment in Subject With Benign Masseteric Hypertrophy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT01-KR17BMH305
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Masseter Muscle Hypertrophy
MeSH Terms: conditions — Masticatory Muscles, Hypertrophy of | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MEDITOXIN (Experimental)
  Interventions: Drug: Meditoxin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Meditoxin — Meditoxin (Botulinum toxin type A)
  Arms: MEDITOXIN
Drug: Placebo — Placebo (Normal saline)
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of MEDITOXIN in subjects with benign masseteric hypertrophy compared with placebo

ELIGIBILITY:
Inclusion Criteria:

* subject who aged 20 to less than 65 years
* subject with benign masseteric hypertrophy

Exclusion Criteria:

* subject not appropriate for participating in this study according to the investigator's opinion
* subject with known an anaphylactic response to BoNT/A and other involved ingredients of Investigational product

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
changes in the thickness of the masseter muscle during maximum clenching measured using ultrasound at week 12 from baseline | 12 week follow-up visit

SECONDARY OUTCOMES:
changes in the thickness of the masseter muscle as usual measured using ultrasound at week 12 from baseline | 12 week follow-up visit

CONTACTS AND LOCATIONS:
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea